CLINICAL TRIAL: NCT04820868
Title: A Blinded Prospective Study on Validation of the Performance of a cfDNA Methylation-based Model for Early Cancer Detection
Brief Title: The Unintrusive Detection of EaRly-stage Cancers
Acronym: THUNDER
Status: Completed | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Guangzhou Burning Rock Dx Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: RSCD2020003
Record Dates: First submitted 2021-03-26; First posted 2021-03-29 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Cancer
Keywords: Cancer; Liquid biopsy; Cell-free DNA (cfDNA); Early detection
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cancer Arm: Participants with new diagnosis of cancer, from whom blood samples will be collected
  Interventions: Device: Multi-cancer early detection test
- Healthy Arm: Participants without known presence of malignancies or benign diseases, from whom blood samples will be collected
  Interventions: Device: Multi-cancer early detection test

INTERVENTIONS:
Device: Multi-cancer early detection test — Blood collection and multi-cancer early detection test

SUMMARY:
According to a previous study, a cell-free DNA (cfDNA) methylation-based model showed high sensitivity and specificity (80.6% and 98.3%) in blood-based multi-cancer detection. In this way, a multi-center, prospective, single-blind study (THUNDER study) is designed to further validate the performance of the cfDNA methylation-based model for early cancer detection. Blood RNA markers will also be evaluated. The study will enroll approximately 2508 participants, including participants with malignancies and healthy participants.

ELIGIBILITY:
Inclusion Criteria for All the Participants:

* Ability to provide a written informed consent
* 40-75 years old
* Ability to comply with study procedures

Exclusion Criteria for All the Participants:

* Pregnancy or lactating women
* Recipients of organ transplant or prior non-autologous (allogeneic) bone marrow transplant or stem cell transplant
* Recipients of blood transfusion within 7 days prior to study blood draw
* Recipients of any anti-cancer therapy within 30 days prior to study blood draw, due to diseases other than cancer

Inclusion Criteria for Cancer Arm Participants:

* Confirmed diagnosis or suspicious cases of cancer within 42 days prior to study blood draw.
* No prior anti-cancer therapy (local or systematic) prior to study blood draw

Exclusion Criteria for Cancer Arm Participants:

* Known prior or current diagnosis of other types of malignancies or multiple primary tumors
* Diagnosis of benign diseases by histopathological assessments
* No confirmed diagnosis of cancer by histopathological or radiological assessments within 42 days of study blood draw, or inability to characterize whether the lesion is malignant or benign
* Non-small-cell lung cancer patients with ground-class nodularity by radiological examination
* Diagnosis of precancerous lesions

Inclusion Criteria for Healthy Arm Participants:

* No cancer-related symptoms or discomfort within 30 days prior to study blood draw
* No clinically significant finding by physical examinations, hematological assessment, urinalysis, LDCT or ultrasound
* No clinically significant finding by breast ultrasound or Molybdenum Target Mammography Detection, or Thinprep cytologic test (TCT) detection for female participants
* No active hepatitis B or hepatitis C infection

Exclusion Criteria for Healthy Arm Participants:

* Prior or ongoing treatment of cancer within 3 years prior to study blood draw
* Clinically significant or uncontrolled comorbidities

Ages: 40 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Eligible participants will be recruited from medical centers and assigned into two arms, including participants with new diagnosis of malignancies and healthy participants.
Sampling Method: Non-Probability Sample
Enrollment: 2508 (Actual)
Dates: Start 2021-04-23 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of early detection of 6 types of cancers and Tissue of origin (TOO) accuracy of a cfDNA methylation-based model | 7 months

SECONDARY OUTCOMES:
Sensitivity, specificity and TOO accuracy of a cfDNA methylation-based model in different stages or pathological types of cancer | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Gao, M.D., Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No